CLINICAL TRIAL: NCT04344054
Title: A Phase II, Observer-blinded, Randomized, Active-controlled Study to Examine the Immunogenicity and Safety of Rotarix® and RV3-BB When Co-administered/Boosted With Trivalent P2-VP8 Subunit Rotavirus Vaccine Candidate in Healthy Infants in South Africa
Brief Title: Mixed Schedule Study of Live Oral Rotavirus Vaccines and Trivalent P2-VP8 Subunit Rotavirus Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: SK Bioscience Co., Ltd. (Industry); Murdoch Childrens Research Institute (Other); Children's Hospital Medical Center, Cincinnati (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVIA 082
Record Dates: First submitted 2020-04-06; First posted 2020-04-14 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Rotavirus Vaccine
Keywords: Parental Rotavirus Vaccine; Rotarix; RV3-BB; TV P2-VP8; Mixed schedule; Rotavirus Booster
MeSH Terms: interventions — RIX4414 vaccine

STUDY DESIGN:
Intervention Model Description: The study will enroll infants in six arms divided into two cohorts enrolling infants at birth (0-6 days) or at approximately 6 weeks of age. Within each cohort, the enrolled infants will be randomized to the three arms in a ratio of 6:6:5.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants will receive vaccine as per the assigned treatment to the arm to which he/she has been randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental): RV3-BB/TV P2-VP8 boost
  Interventions: Biological: RV3-BB; Biological: Trivalent P2-VP8 Booster dose
- Arm 2 (Experimental): RV3-BB/TV P2-VP8 co-administered
  Interventions: Biological: RV3-BB; Biological: Trivalent P2-VP8
- Arm 3 (Experimental): RV3-BB primed TV P2-VP8
  Interventions: Biological: Trivalent P2-VP8; Biological: RV3-BB birth dose
- Arm 4 (Experimental): Rotarix®/TV P2-VP8 Boost
  Interventions: Biological: Rotarix; Biological: Trivalent P2-VP8 Booster dose
- Arm 5 (Experimental): Rotarix®/TV P2-VP8 co-administered
  Interventions: Biological: Trivalent P2-VP8; Biological: Rotarix
- Arm 6 (Experimental): TV P2-VP8 alone
  Interventions: Biological: Trivalent P2-VP8

INTERVENTIONS:
Biological: RV3-BB — 1.0 mL of the thawed rotavirus vaccine to be administered orally at birth, 6 weeks and 10 weeks of age
  Arms: Arm 1; Arm 2
Biological: Trivalent P2-VP8 — 0.5 mL of vaccine containing 90 μg of the TV P2-VP8 antigen; IM; at approximately 6, 10 and 14 weeks of age
  Arms: Arm 2; Arm 3; Arm 5; Arm 6
Biological: Rotarix — 1.5 mL of the liquid vaccine containing the RIX4414 strain of human rotavirus vaccine to be administered orally at 6 weeks and 10 weeks of age.
  Arms: Arm 4; Arm 5
Biological: RV3-BB birth dose — 1.0 mL of the thawed rotavirus vaccine to be administered orally at birth.
  Arms: Arm 3
Biological: Trivalent P2-VP8 Booster dose — 0.5 mL of vaccine containing 90 μg of the TV P2-VP8 antigen; IM; at 14 weeks of age
  Arms: Arm 1; Arm 4

SUMMARY:
The study will evaluate safety and immunogenicity of LORV (Rotarix and RV3-BB) when TV P2-VP8, a parentally administered rotavirus vaccine is administered either concomitantly or as a prime/boost model. Participants would be newborn babies or infants approximately at 6 weeks of age ta the time of enrollment. The vaccines will be administered at birth (only for one cohort) and at 6, 10 and 14 weeks. Immune response will be assessed prior to first vaccination, 14 weeks and at 18 weeks of age. The study will also evaluate the shedding of Rotarix virus after a challenge dose administered 28 days after last investigational product administration. Safety assessments will be conducted throughout the study duration.

DETAILED DESCRIPTION:
This is a phase II, observer-blinded, multi-center, randomized and active-controlled study enrolling healthy infants 0-6 days of age or 6-8 weeks of age. The study will enroll infants in six arms divided into two cohorts enrolling infants at birth (0-6 days) and approximately 6 weeks of age. Within each cohort, the enrolled infants will be randomized to the three arms in a ratio of 6:6:5. Participants in Cohort A will receive: RV3-BB/TV P2-VP8 boost (arm 1); RV3-BB/TV P2-VP8 co-administered (arm 2); RV3-BB primed TV P2-VP8 (arm 3), while participants in Cohort B will receive: Rotarix®/TV P2-VP8 Boost (arm 4); Rotarix®/TV P2-VP8 co-administered (arm 5); or TV P2-VP8 alone (arm 6). Rotarix® and RV3-BB will be administered orally whereas TV P2-VP8 will be administered intramuscularly. The study will be conducted as an observer-blinded study wherein the treatment assignment within a cohort will be blinded, although allocation to a cohort will be unblinded due to the difference in age at enrolment between the two cohorts. Participants will receive a dose of injectable or oral placebo to maintain blinding.

A blood sample will be obtained from all the participating infants pre-vaccination and post-vaccination at week 14 and week 18 in both cohorts. All serum samples will be tested for serum IgA binding antibody by ELISA using virus lysates prepared from RV3-BB and 89-12 strains. Additionally, anti-P2-VP8 IgG binding and serum neutralizing antibody levels to each of the 3 strains of rotavirus from which TV P2-VP8 is derived will be determined.

Vaccine safety will be evaluated by 1) recording the immediate adverse events for 30 minutes after immunization, 2) solicited adverse events for 7 days after each study vaccination, 3) unsolicited events for 28 days after each dose, and 4) serious adverse events 28 days after last dose of study vaccination.

All participants in all the study arms will receive a challenge dose of Rotarix® at visit 5following completion of primary series of vaccinations. Stool sample will be collected to evaluate vaccine viral shedding.

The primary objective of the study is to compare the immunogenicity in participants receiving LORV co-administration with TV P2- VP8 or those receiving the TV P2-VP8 booster after receiving a standalone LORV primary series with the standalone LORV. A comparison of immune responses to birth dose of RV3-BB boosted with TV P2-VP8 to TV P2-VP8 administered alone will also be conducted. All primary immunogenicity analysis will be based on LORV specific serum anti-rotavirus IgA antibody concentration. Placebo administration (oral and parenteral) were appropriately placed to facilitate blinding.

The secondary objective were to compare the different treatment regimens within a cohort using serum anti-P2-VP8 IgG antibodies and neutralizing antibodies to each of the 3 strains of rotavirus from which TV P2-VP8 is derived.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female infants as established by medical history and clinical examination at enrollment.
2. Age: ≤ 6 days old (Cohort A) or between the age of 6-8 weeks (42-56 days; inclusive) (Cohort B)
3. Birth weight of ≥ 2500 grams.
4. Parent's/legally acceptable representative's (LAR) ability and willingness to provide informed consent.
5. Parent/LAR confirms intention to stay in the area and bring their infant for the required study visits.

Exclusion Criteria:

1. Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrollment; temporary exclusion.
2. Presence of acute disease at the time of enrollment; temporary exclusion.
3. Presence of fever on the day of enrollment (axillary temperature ≥37.5 °C); temporary exclusion.
4. Concurrent participation in another clinical trial throughout the entire timeframe of this study.
5. Presence of any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would compromise the child's health or is likely to result in non-conformance to the protocol.
6. History of premature birth (<37 weeks gestation) as per the investigator's assessment.
7. History of congenital abdominal disorders, intussusception, abdominal surgery.
8. Known or suspected impairment of immunological function based on medical history and physical examination.
9. Prior receipt of or intent to receive age specified EPI vaccines including rotavirus vaccine, outside of the study center and during study participation.
10. A known sensitivity or allergy to any components of the study medication.
11. Clinically detectable congenital anomaly or genetic defect.
12. History of persistent diarrhea (defined as diarrhea more than 14 days). Not applicable for selection of Cohort A.
13. Participant's parent/LAR not able, available or willing to accept active follow-up by the study staff.
14. Receipt of any immunoglobulin therapy and/or blood products since birth or planned administration during the study period.
15. History of chronic administration (defined as more than 14 days) of high doses of immunosuppressant including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study. Not applicable for selection of Cohort A.
16. Any medical condition in the parents/infants that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parent's/LAR's ability to give informed consent.

Max Age: 56 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 850 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity 1 | 4 weeks after the last vaccination within each regimen being compared.
  Immunogenicity: Between-arm comparisons (all comparisons except for LORV alone vs TV P2-VP8-boosted LORV) will be performed by computing Geometric Mean Concentration (GMC) ratios for LORV-specific serum anti-rotavirus IgA antibody and corresponding confidence intervals.
Immunogenicity 2 | 4 weeks after completion of LORV (Week 14)
  Immunogenicity: Within-arm evaluation of boosting will be performed using the geometric mean fold rise (GMFR) of LORV-specific serum anti-rotavirus IgA antibody and its corresponding confidence interval.
Immunogenicity 3 | 4 weeks post-boost (Week 18)
  Immunogenicity: Within-arm evaluation of boosting will be performed using the geometric mean fold rise (GMFR) of LORV-specific serum antirotavirus IgA antibody and its corresponding confidence interval.
Safety 1: Percentage of participants reporting immediate adverse events after each vaccination | within 30 minutes' post-vaccination
  Immediate Adverse Events: Percentage of participants reporting immediate adverse events after each vaccination
Safety 2: Percentage of participants reporting solicited post-vaccination reactogenicity | 7 day period after each vaccination
  Solicited Adverse Events: Percentage of participants reporting solicited post-vaccination reactogenicity
Safety 3: Percentage of participants reporting unsolicited AEs | from first vaccination through 4 weeks after the last vaccination
  Unsolicited Adverse Events: Percentage of participants reporting unsolicited AEs
Safety 4: Percentage of participants reporting SAEs | from first vaccination through 4 weeks after the last vaccination of each study participant
  Serious Adverse Events: Percentage of participants reporting SAEs

SECONDARY OUTCOMES:
Immunogenicity 1 | 4 weeks after the last vaccination within each regimen being compared
  Between- and within-arm comparisons for serum IgA will be performed using GMC ratios and GMFRs, respectively
Immunogenicity 2 | 4 weeks after the last vaccination
  Seroconversion rate for anti-rotavirus IgA antibodies.
Immunogenicity 3 | 4 weeks after the last vaccination
  Seropositivity rate for anti-rotavirus IgA antibodies.
Immunogenicity 4 | 4 weeks after the last vaccination
  Seroresponse rate for anti-rotavirus IgA antibodies.
Immunogenicity 5 | 4 weeks after the last vaccination
  Geometric Mean Concentration (GMC) ratios and Geometric Mean Fold Rise (GMFR) for serum anti-P2-VP8 IgG antibodies.
Immunogenicity 6 | 4 weeks after the last vaccination
  Seroresponse rate for serum anti-P2-VP8 IgG antibodies.
Immunogenicity 7 | 4 weeks after the last vaccination
  Geometric Mean Titers (GMT) ratios and Geometric Mean Fold Rise (GMFR) of TV P2-VP8-specific serum neutralizing antibodies.
Immunogenicity 8 | 4 weeks after the last vaccination
  Seroresponse rate of TV P2-VP8-specific serum neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cryz, PhD, Study Director — PATH
Locations (2):
- South Africa (2):
  - Wits RHI Shandukani Research Centre, Johannesburg, Gauteng
  - Vaccine and Infectious Diseases Analytics (VIDA) - formerly known as Respiratory and Meningococcal Pathogens Research Unit (RMPRU), Johannesburg, Gauteng

IPD SHARING:
Plan to Share IPD: Yes
Summary results for primary and secondary objectives to be posted at CT.gov.
Supporting Information: Study Protocol
Time Frame: Within 12 months of completion of study
Access Criteria: Researchers who provide a methodologically sound proposal may be provided access after sponsor permission.